CLINICAL TRIAL: NCT05614219
Title: Can Biochemistry Interpretive Comments on Elevated Cholesterol Levels, Increase Referrals to Lipid Clinics and Detection Rate of Familial Hypercholesterolemia? A Step Wedge Cluster Randomized Controlled Trial.
Brief Title: Familial Hypercholesterolemia Interpretive Comment - Nudging to Detection.
Acronym: FIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Knold, MD, Odense University Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: FINDRSYD22
Record Dates: First submitted 2022-10-27; First posted 2022-11-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Familial Hypercholesterolemia
Keywords: Familial Hypercholesterolemia; Biochemistry interpretive comment; Low-density lipoprotein cholesterol levels; Screening
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: Step wedge cluster randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biochemistry interpretive comment on LDL-C levels (Experimental): The general practitioners and hospital wards will be allocated in cluster according to their providing lab, and stepwise implement the comment on LDL-C > 4 mmol/L in persons under the age of 40 and over 5 mmol/L in persons over the age of 40 years. Raising awareness on familial hypercholesterolemia an encouraging to referral.
  Cluster 1. Will from the 01.12.2022 implement comment on LDL-C Cluster 2. Will from the 01.03.2023 implement comment on LDL-C Cluster 3. Will from the 01.06.2023 implement comment on LDL-C Cluster 4.Will from the 01.09.2023 implement comment on LDL-C
  Interventions: Other: Biochemistry interpretive comment on elevated LDL-C levels
- Control (No Intervention): The clusters will act as their own controls, due to the stepwise implementation of the comment.
  Cluster 2: Will not implement the comment before the 01.03.2023 Cluster 3: Will not implement the comment before the 01.06.2023 Cluster 4: Will not implement the comment before the 01.09.2023

INTERVENTIONS:
Other: Biochemistry interpretive comment on elevated LDL-C levels — The interpretive comment on LDL-C will encourage for excluding secondary dyslipidemia (measuring Hba1C, TSH and checking current drugs and talk about diet). If secondary dyslipidemia ca be excluded we encourage to referral to lipid clinic. Familial hypercholesterolemia should be suspected if LDL-C > 4 mmol/L in persons under the age of 40, or LDL-C > 5 mmol/L in persons over the age of 40. The biochemistry interpretive comment will thus be released to the referring physician if the blood sample meet the criteria above. We advice that in pregnant women to control elevated LDL-C after childbirth.
  Arms: Biochemistry interpretive comment on LDL-C levels

SUMMARY:
Familial hypercholesterolemia is the most common inherited disease of the lipid metabolism, however it remains underdiagnosed. Only 15 % of 30.000 possible patients have been found in Denmark. This quality assessing project will through a step wedge cluster randomized controlled trial evaluate establishment of a biochemistry interpretive comment on elevated LDL-C levels. The study will test if the comment results in an increase in referred patients to the lipid clinics of Southern Denmark as the primary endpoint, and as the secondary endpoint in more patients diagnosed with familial hypercholesterolemia. The project will run in totally 52 weeks and will in steps initiate the comment from the different laboratories in the Region of Southern Denmark.

DETAILED DESCRIPTION:
Introduction:

Familial hypercholesterolemia (FH) is the most common inherited disease of the lipid metabolism with a prevalence of approximately 1/200. It is estimated that only 15 % of the estimated 30.000 patients in Denmark has been diagnosed. With high risk of atherosclerotic coronary disease, it is estimated that there is a great potential regarding cardiovascular health and health economics by early initiation of lipid lowering treatment and cascade screening of families.

All doctors can refer to lipid clinics on the suspicion of FH. FH should be suspected when low-density lipoprotein - cholesterol (LDL-C) is extremely elevated without any other explanation in young individuals, or in families with premature cardiovascular disease. The diagnosis is made from clinical scoring systems as the Simon Broome criteria, Dutch Lipid Clinical Network criteria and the MEDPED criteria including genetic test. The treatment is lipid-lowering drugs including statins, ezetimibe and PCSK9-inhibitor in case of insufficient effect.

In the last 12-14 years systematic cascade screening of FH families have been used in Denmark to track and find FH patients. The patients have since 2020 been registered in the National clinical quality database for FH.

However FH remains an under diagnosed disease, resulting in premature ischemic cardiovascular disease and premature cardiovascular death. Thus, there is a need for optimized screening for FH and more projects are already initiated.

Detecting more FH patients will demand an increased attention on elevated cholesterol. A biochemistry interpretive comment on elevated LDL-C according to the Danish FH Guideline regarding when to suspect FH, encouraging to further investigation for secondary dyslipidemia and successive referral to lipid clinic suspecting FH, can theoretically increase the awareness of FH. In England a survey has shown that general practitioners ask for interpretive comments on biochemistry analyses and 19 % of the general practitioners demands a comment on the lipid analyses.

A minor case control study in Australia have shown that interpretive comment on lipid profiles led to a significant reduction in LDL-C compared to controls, and increased the rate of referral by 11.5 % in cases compared to 1 % in controls, however only a minority was referred. The study was relatively small with 96 cases and 100 controls and an interpretive comment was activated when LDL-C > 6.5 mmol/L. However, the study is supported by a prospective case control study by the same research group including 231 patients with LDL-C > 6.5 mmol/L, where all doctors received an interpretive comment on elevated the LDL-C, raising suspicion to FH, but only cases received a comment which encouraged to referral to lipid clinic. Hereby 18 % of cases was referred compared to 8 % of controls. This indicates that in a minor population in another country, establishment of an interpretive comment on LDL-C could increase referral rate by 10 %. The prospective case control study concludes that the interpretive comment increases the detection rate of FH patients.

We want to evaluate implementation of an interpretive comment on elevated LDL-C levels in the Region of Southern Denmark. Compared to the Australian studies we expect to get more referrals since our cut-off for referral is lower (LDL-C 4 or 5 mmol/L depending on age). A strength in our study is the prospective step wedge RCT design.

Purpose and scientifically question:

This study will try to optimize screening for FH by investigating the effect of a biochemistry interpretive comment when LDL-C is significantly elevated according to the Danish FH guideline. The comment will encourage to further investigation and referral to local lipid clinic. The purpose is to test the effect of the interpretive comment regarding the proportion of patients referred to the lipid clinics as the primary endpoint. As the secondary endpoints we wish to calculate the change in LDL-C from referral to first contact in the lipid clinic, and the proportion of new diagnosed patients with FH at the lipid clinics in the Region of Southern Denmark.

This study will evaluate if it is possible to receive more referrals to the lipid clinics and find more patients with FH by an interpretive comment on cholesterol levels, encouraging to investigate for secondary dyslipidemia, and successive refer to lipid clinic in case of no explanation of the elevated LDL-C. The study will elucidate how many patients we have to refer, to find one patient with FH?

Method and material:

This study will through a step wedge cluster randomized controlled trial, investigate if establishment of the interpretive comment will result in more referrals and as the primary endpoint in more diagnosed patients with FH in the Region of Southern Denmark.

The material will consist of referred patients to the lipid clinics of Southern Denmark. The general practitioners and medical wards in the Region of Southern Denmark will be allocated in clusters according to the providing lab, totally 4 clusters. The clusters will be randomised to stepwise implementation of the biochemistry interpretive comment on cholesterol samples meeting the following criteria. FH should be suspected if LDL-C > 4 mmol/L in persons under the age of 40, or LDL-C > 5 mmol/L in persons over the age of 40 according to the Danish guideline on FH. Randomization will be dobbeltblinded to data analyzing researchers and the general practitioners and wards receiving the interpretive comment.

The clusters will act as their own controls, the intervention being the biochemistry interpretive comment. The first cluster will implement the comment from the 01.12.2022 and after 12 weeks the next cluster will implement the comment. After 48 weeks all clusters will have implemented the interpretive comment. Further 8 weeks will act as buffer resulting in a totally study period of 52 weeks.

The Study will elucidate the proportion of referred patients and patients diagnosed with FH in the Region of Southern Denmark, after implementation of the interpretive comment.

The study will elucidate whether the proportion of referrals and diagnosed patients increases after implementation of the interpretive comment in the specific cluster or between the clusters.

The proportion of referred patients will be registered through data from the electronic patient journal system (EPJ). The reffered patients will be stratified both geographically and according to the referring physicians electronic laboratory system to account for bias regarding how the interpretive comment appears in the different systems, and whether this influence referral rate. The proportion of patients diagnosed with FH will be registered through ICD-10 codes in EPJ and crosschecked with Dutch Lipid Clinical score from the patient journal, including lipid profile and genetics to ensure a valid diagnosis. Furthermore HbA1c, TSH, liver- and kidney parameters and lipid profile will be registered as patient baseline characteristic to exclude patients with secondary dyslipidemia and to follow changes in LDL-C from referral to first lipid clinic contact. The study will furthermore elucidate how many patients there need to be referred to find one patient with FH.

Ethics

There is no need for information on an individual level, because the study is focusing on an organizational level as a step wedge cluster design. The patients can always deny further investigation or referral, and in this study we do not encourage to take blood samples without clinical indication. Instead we encourage through the biochemistry interpretive comment to act on blood samples already taken. The scientifically committee of Southern Denmark finds no indication for registration of the study because it is a study of assessing quality (Record number. S-20222000-106). The study will be registered in the Region of Southern Denmarks list of Research projects.

ELIGIBILITY:
Inclusion Criteria:

* All referred patients to the lipid clinics of Southern Denmark
* LDL-C < 4 mmol/L in persons under the age of 40.
* LDL-C > 5 mmol/L in persons over the age of 40.

Exclusion Criteria:

Pregnancy and Secondary dyslipidemia

* Dysregulated diabetes. Hba1C < 48
* Dysregulated hypothyreosis. Elevated TSH.
* Kombined hyperlipidiemia TG > 4 mmol/L
* Nefrotic syndrome: proteinuria > 3 g/L and s-albumin < 30 g/l
* Cholestasis (alcalic fosfatase > 105 U/L and GGT > 55 U/L) 14 days prior to LDL-C measuring
* Pharmacological induced hyperlipidimia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients reffered to lipid clinic | 12-18 months
  Proportion of referred patients to lipid clinics in the region of Southern Denmark after establishment of interpretive comment on LDL-C, compared to proportion before the comment.
Diagnosed patients with Familial Hyperchoelsterolemia | During 9-12 months due to waiting time for genetic test
  Proportion of patients diagnosed with familial hypercholesterolemia (Dutch clinical lipid score > 8) in the Region of Southern Denmark after establishment of interpretive comment on LDL-C, compared to proportion before the comment.

SECONDARY OUTCOMES:
Change in LDL-C | 3-6 months
  Change in LDL-C levels from referral to first contact in lipid clinic
Familial hypercholesterolemia mutations | 9-12 months due to waiting time for genetic test
  Number of genetic test with mutations related to familial hypercholesterolemia
Hba1C | 3 months
  Mean Hba1C at referral as baseline value
TSH | 3 months
  Mean TSH at referral as baseline value
Triglycerides | 3 months
  Mean triglycerides at referral as baseline value and change in triglycerides at first visit in lipid clinic.
HDL-Cholesterol | 3 months
  Mean HDL-Cholesterol at referral as baseline value and change in HDL-Cholesterol at first visit in lipid clinic.
Lipoprotein(a) | 3 months
  Mean Lipoprotein(a) as a baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Finn Lund Henriksen, Ph.d., Principal Investigator — Departement of Cardiology, Odense University Hospital
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense, Funen
  - Departement of Cardiology, Odense University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: No
The results will be published and shared in an international peer reviewed journal.

REFERENCES:
- [Background] Levenson AE, de Ferranti SD. Familial Hypercholesterolemia. In: Feingold KR, Anawalt B, Boyce A, Chrousos G, de Herder WW, Dhatariya K, et al., editors. Endotext. South Dartmouth (MA)2000.
- [Background] Bundgaard H SMea. Regionernes klinisk kvalitetsdatabase. Familiær hyperkolesterolæmi databasen. 2020 [Available from: https://www.rkkp.dk/kvalitetsdatabaser/databaser/databasen-for-familiaer-hyperkolesterolaemi/
- [Background] Rosso A, Pitini E, D'Andrea E, Massimi A, De Vito C, Marzuillo C, Villari P. The Cost-effectiveness of Genetic Screening for Familial Hypercholesterolemia: a Systematic Review. Ann Ig. 2017 Sep-Oct;29(5):464-480. doi: 10.7416/ai.2017.2178. PMID 28715059
- [Background] Sturm AC, Knowles JW, Gidding SS, Ahmad ZS, Ahmed CD, Ballantyne CM, Baum SJ, Bourbon M, Carrie A, Cuchel M, de Ferranti SD, Defesche JC, Freiberger T, Hershberger RE, Hovingh GK, Karayan L, Kastelein JJP, Kindt I, Lane SR, Leigh SE, Linton MF, Mata P, Neal WA, Nordestgaard BG, Santos RD, Harada-Shiba M, Sijbrands EJ, Stitziel NO, Yamashita S, Wilemon KA, Ledbetter DH, Rader DJ; Convened by the Familial Hypercholesterolemia Foundation. Clinical Genetic Testing for Familial Hypercholesterolemia: JACC Scientific Expert Panel. J Am Coll Cardiol. 2018 Aug 7;72(6):662-680. doi: 10.1016/j.jacc.2018.05.044. PMID 30071997
- [Background] Raal FJ, Hovingh GK, Catapano AL. Familial hypercholesterolemia treatments: Guidelines and new therapies. Atherosclerosis. 2018 Oct;277:483-492. doi: 10.1016/j.atherosclerosis.2018.06.859. PMID 30270089
- [Background] Hedegaard BS. A danish nationwide study og individuals suspected of FH referred from general practice to lipid clinics: Clinical characteristics, plasma lpipoprotein(A) and final diagnosis. Atherosclerosis. 2021.
- [Background] Schmidt EB, Hedegaard BS, Retterstol K. Familial hypercholesterolaemia: history, diagnosis, screening, management and challenges. Heart. 2020 Dec;106(24):1940-1946. doi: 10.1136/heartjnl-2019-316276. Epub 2020 Sep 15. No abstract available. PMID 32933999
- [Background] Schmidt EB, Henriksen FL, Kanstrup HL. Familiær hyperkolesterolæmi holdningspapir Dansk Cardiologisk Selskab2019 [08.04. 2022]. Available from: https://nbv.cardio.dk/media/com_reditem/files/customfield/item/7349/601670e648780b94c9cf26375caef524dcdb2270.pdf
- [Background] Barlow IM. Are biochemistry interpretative comments helpful? Results of a general practitioner and nurse practitioner survey. Ann Clin Biochem. 2008 Jan;45(Pt 1):88-90. doi: 10.1258/acb.2007.007134. PMID 18275680
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947